CLINICAL TRIAL: NCT03783195
Title: Genetic-specific Effects of Fructose on Liver Lipogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-3348; P30DK056336-16S1 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-05

CONDITIONS: NAFLD
Keywords: Glucose; Fructose; Fatty-liver; Polymorphisms; Imaging; Fibroscan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Intervention Model Description: Participants are assigned to high genetic risk score group in parallel to low genetic risk score group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High GRS group (Experimental): This group consists of individuals who are in the highest quartile of the genetic risk score (GRS) and will ingest one sugar drink (equal to 2 soft drinks) per day for 3 weeks. The GRS is computed by adding the number of alleles that increase the risk for liver lipogenesis or fatty liver.
  Interventions: Other: Sugar drink
- Low GRS group (Experimental): This groups consists of individuals who are in the lowest quartile of the genetic risk score (GRS) and will ingest one sugar drink (equal to 2 soft drinks) per day for 3 weeks. The GRS is computed by adding the number of alleles that increase the risk for liver lipogenesis or fatty liver.
  Interventions: Other: Sugar drink

INTERVENTIONS:
Other: Sugar drink — A sugar drink made with 1.2 g/kg body weight of added sugar( 0.75g/kg body weight of fructose + 0.45g/kg body weight of glucose) and 24oz water

SUMMARY:
The primary goal of this study is to identify a set of genotypes that increase the risk for nonalcoholic fatty liver disease (NAFLD) and predispose individuals to increased de novo lipogenesis (DNL) and liver fat accumulation when exposed to fructose intake. The proposed goal will be achieved through the completion of following aims:

1. To determine the impact of prolonged exposure of fructose on hepatic lipid accumulation in Caucasian individuals with high and low genetic risk for NAFLD,
2. to determine the impact of acute exposure of fructose on hepatic DNL, and
3. to determine the relationship between markers of DNL, liver fat accumulation and serum concentrations of lipids, uric acid and liver function markers before and after the fructose challenge.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Non-alcoholic fatty liver disease (NAFLD) is characterized by fat accumulation in liver cells not caused by alcohol. A leading cause of chronic liver disease in the US, NAFLD represents a group of disorders including steatosis, nonalcoholic steatohepatitis with fibrosis. It has substantially risen in prevalence over the last two decades with the estimated prevalence being 20% among US adults and 25% in young adults (18-39 years). Over 64 million individuals are believed to have NAFLD with annual medical costs rising to more $100 billion. More common in individuals who are obese or diabetic and/or have metabolic syndrome, NAFLD has been associated with increased cirrhosis, liver-related mortality and hepatocellular carcinoma.

Both genetic and environmental, including nutritional, factors contribute to the onset and progression of NAFLD. Increased consumption of sugar-sweetened, fructose-rich beverages has been linked to NAFLD. Fructose, commonly found in soft drinks, fruit juices and energy drinks, affects many metabolic processes, foremost being an increase in fat accumulation in the liver and hence, NAFLD. Genome-wide and candidate gene studies have identified several genes associated with NAFLD. However, none of these studies have shown the cumulative effects of single nucleotide polymorphisms (SNPs) on changes in liver fat when exposed to fructose. The results from this study can be extrapolated to larger cohorts and other ethnicities and are therefore, expected to lay the foundation for developing personalized nutritional plans.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 12 - 40 years
2. No history of alcohol abuse (> 7 drinks per week)
3. History of fructose intake of < 14 drinks per week
4. Caucasian ethnicity
5. BMI > 25kg/m² - 32kg/m² or 85th -99th percentile but otherwise healthy

Exclusion Criteria:

1. ages < 12 and > 40 years
2. Pregnant/lactating
3. known alcohol abuse or fructose intake > 14 drinks per week
4. not of Caucasian ethnicity
5. glucose levels > 100 mg/dL if fasting, > 140mg/dL if within 2 hours post meal and > 200 mg/dL if random sample
6. taking anti-hypertensive, anti-diabetic, uric acid and/or lipid-lowering medications
7. known diagnosis of diabetes, fructose intolerance, chronic kidney disease, NAFLD or any liver-related disease, hypertriglyceridemia, polycystic ovary syndrome, hypothyroidism, obstructive sleep apnea, hypopituitarism and hypogonadism
8. BMI < 25kg/m² or > 32 kg/m² or < 85th or > 99th percentile
9. Liver fat fraction >5% as per baseline MRI scan

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroja Voruganti, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Supporting Information: Study Protocol
Time Frame: 9- 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by the institutional review board, independent ethics committee or research ethics committee, as applicable and an executed data use agreement with UNC.

REFERENCES:
- [Background] Younossi ZM, Blissett D, Blissett R, Henry L, Stepanova M, Younossi Y, Racila A, Hunt S, Beckerman R. The economic and clinical burden of nonalcoholic fatty liver disease in the United States and Europe. Hepatology. 2016 Nov;64(5):1577-1586. doi: 10.1002/hep.28785. Epub 2016 Sep 26. PMID 27543837
- [Background] Vos MB, Kimmons JE, Gillespie C, Welsh J, Blanck HM. Dietary fructose consumption among US children and adults: the Third National Health and Nutrition Examination Survey. Medscape J Med. 2008 Jul 9;10(7):160. PMID 18769702
- [Background] Moore JB, Gunn PJ, Fielding BA. The role of dietary sugars and de novo lipogenesis in non-alcoholic fatty liver disease. Nutrients. 2014 Dec 10;6(12):5679-703. doi: 10.3390/nu6125679. PMID 25514388
- [Background] Faeh D, Minehira K, Schwarz JM, Periasamy R, Park S, Tappy L. Effect of fructose overfeeding and fish oil administration on hepatic de novo lipogenesis and insulin sensitivity in healthy men. Diabetes. 2005 Jul;54(7):1907-13. doi: 10.2337/diabetes.54.7.1907. PMID 15983189
- [Background] Alwahsh SM, Gebhardt R. Dietary fructose as a risk factor for non-alcoholic fatty liver disease (NAFLD). Arch Toxicol. 2017 Apr;91(4):1545-1563. doi: 10.1007/s00204-016-1892-7. Epub 2016 Dec 19. PMID 27995280
- [Background] Stanhope KL, Schwarz JM, Keim NL, Griffen SC, Bremer AA, Graham JL, Hatcher B, Cox CL, Dyachenko A, Zhang W, McGahan JP, Seibert A, Krauss RM, Chiu S, Schaefer EJ, Ai M, Otokozawa S, Nakajima K, Nakano T, Beysen C, Hellerstein MK, Berglund L, Havel PJ. Consuming fructose-sweetened, not glucose-sweetened, beverages increases visceral adiposity and lipids and decreases insulin sensitivity in overweight/obese humans. J Clin Invest. 2009 May;119(5):1322-34. doi: 10.1172/JCI37385. Epub 2009 Apr 20. PMID 19381015
- [Background] Stanhope KL, Medici V, Bremer AA, Lee V, Lam HD, Nunez MV, Chen GX, Keim NL, Havel PJ. A dose-response study of consuming high-fructose corn syrup-sweetened beverages on lipid/lipoprotein risk factors for cardiovascular disease in young adults. Am J Clin Nutr. 2015 Jun;101(6):1144-54. doi: 10.3945/ajcn.114.100461. Epub 2015 Apr 22. PMID 25904601
- [Background] Softic S, Gupta MK, Wang GX, Fujisaka S, O'Neill BT, Rao TN, Willoughby J, Harbison C, Fitzgerald K, Ilkayeva O, Newgard CB, Cohen DE, Kahn CR. Divergent effects of glucose and fructose on hepatic lipogenesis and insulin signaling. J Clin Invest. 2017 Nov 1;127(11):4059-4074. doi: 10.1172/JCI94585. Epub 2017 Oct 3. PMID 28972537
- [Background] Basaranoglu M, Basaranoglu G, Bugianesi E. Carbohydrate intake and nonalcoholic fatty liver disease: fructose as a weapon of mass destruction. Hepatobiliary Surg Nutr. 2015 Apr;4(2):109-16. doi: 10.3978/j.issn.2304-3881.2014.11.05. PMID 26005677
- [Background] Johnson RJ, Nakagawa T, Sanchez-Lozada LG, Shafiu M, Sundaram S, Le M, Ishimoto T, Sautin YY, Lanaspa MA. Sugar, uric acid, and the etiology of diabetes and obesity. Diabetes. 2013 Oct;62(10):3307-15. doi: 10.2337/db12-1814. PMID 24065788
- [Background] Zhou Y, Wei F, Fan Y. High serum uric acid and risk of nonalcoholic fatty liver disease: A systematic review and meta-analysis. Clin Biochem. 2016 May;49(7-8):636-42. doi: 10.1016/j.clinbiochem.2015.12.010. Epub 2015 Dec 29. PMID 26738417
- [Background] Goran MI, Walker R, Allayee H. Genetic-related and carbohydrate-related factors affecting liver fat accumulation. Curr Opin Clin Nutr Metab Care. 2012 Jul;15(4):392-6. doi: 10.1097/MCO.0b013e3283544477. PMID 22617559
- [Background] Speliotes EK, Yerges-Armstrong LM, Wu J, Hernaez R, Kim LJ, Palmer CD, Gudnason V, Eiriksdottir G, Garcia ME, Launer LJ, Nalls MA, Clark JM, Mitchell BD, Shuldiner AR, Butler JL, Tomas M, Hoffmann U, Hwang SJ, Massaro JM, O'Donnell CJ, Sahani DV, Salomaa V, Schadt EE, Schwartz SM, Siscovick DS; NASH CRN; GIANT Consortium; MAGIC Investigators; Voight BF, Carr JJ, Feitosa MF, Harris TB, Fox CS, Smith AV, Kao WH, Hirschhorn JN, Borecki IB; GOLD Consortium. Genome-wide association analysis identifies variants associated with nonalcoholic fatty liver disease that have distinct effects on metabolic traits. PLoS Genet. 2011 Mar;7(3):e1001324. doi: 10.1371/journal.pgen.1001324. Epub 2011 Mar 10. PMID 21423719
- [Background] Davis JN, Le KA, Walker RW, Vikman S, Spruijt-Metz D, Weigensberg MJ, Allayee H, Goran MI. Increased hepatic fat in overweight Hispanic youth influenced by interaction between genetic variation in PNPLA3 and high dietary carbohydrate and sugar consumption. Am J Clin Nutr. 2010 Dec;92(6):1522-7. doi: 10.3945/ajcn.2010.30185. Epub 2010 Oct 20. PMID 20962157
- [Background] Santoro N, Caprio S, Pierpont B, Van Name M, Savoye M, Parks EJ. Hepatic De Novo Lipogenesis in Obese Youth Is Modulated by a Common Variant in the GCKR Gene. J Clin Endocrinol Metab. 2015 Aug;100(8):E1125-32. doi: 10.1210/jc.2015-1587. Epub 2015 Jun 4. PMID 26043229
- [Background] Ter Horst KW, Schene MR, Holman R, Romijn JA, Serlie MJ. Effect of fructose consumption on insulin sensitivity in nondiabetic subjects: a systematic review and meta-analysis of diet-intervention trials. Am J Clin Nutr. 2016 Dec;104(6):1562-1576. doi: 10.3945/ajcn.116.137786. Epub 2016 Nov 9. PMID 27935520
- [Background] Schwarz JM, Noworolski SM, Erkin-Cakmak A, Korn NJ, Wen MJ, Tai VW, Jones GM, Palii SP, Velasco-Alin M, Pan K, Patterson BW, Gugliucci A, Lustig RH, Mulligan K. Effects of Dietary Fructose Restriction on Liver Fat, De Novo Lipogenesis, and Insulin Kinetics in Children With Obesity. Gastroenterology. 2017 Sep;153(3):743-752. doi: 10.1053/j.gastro.2017.05.043. Epub 2017 Jun 1. PMID 28579536
- [Background] Stanhope KL, Bremer AA, Medici V, Nakajima K, Ito Y, Nakano T, Chen G, Fong TH, Lee V, Menorca RI, Keim NL, Havel PJ. Consumption of fructose and high fructose corn syrup increase postprandial triglycerides, LDL-cholesterol, and apolipoprotein-B in young men and women. J Clin Endocrinol Metab. 2011 Oct;96(10):E1596-605. doi: 10.1210/jc.2011-1251. Epub 2011 Aug 17. PMID 21849529
- [Background] Schwarz JM, Noworolski SM, Wen MJ, Dyachenko A, Prior JL, Weinberg ME, Herraiz LA, Tai VW, Bergeron N, Bersot TP, Rao MN, Schambelan M, Mulligan K. Effect of a High-Fructose Weight-Maintaining Diet on Lipogenesis and Liver Fat. J Clin Endocrinol Metab. 2015 Jun;100(6):2434-42. doi: 10.1210/jc.2014-3678. Epub 2015 Mar 31. PMID 25825943
- [Background] Ventura EE, Davis JN, Goran MI. Sugar content of popular sweetened beverages based on objective laboratory analysis: focus on fructose content. Obesity (Silver Spring). 2011 Apr;19(4):868-74. doi: 10.1038/oby.2010.255. Epub 2010 Oct 14. PMID 20948525
- [Background] Akhavan T, Anderson GH. Effects of glucose-to-fructose ratios in solutions on subjective satiety, food intake, and satiety hormones in young men. Am J Clin Nutr. 2007 Nov;86(5):1354-63. doi: 10.1093/ajcn/86.5.1354. PMID 17991646
- [Background] Faix D, Neese R, Kletke C, Wolden S, Cesar D, Coutlangus M, Shackleton CH, Hellerstein MK. Quantification of menstrual and diurnal periodicities in rates of cholesterol and fat synthesis in humans. J Lipid Res. 1993 Dec;34(12):2063-75. PMID 8301227
- [Background] Hudgins LC, Parker TS, Levine DM, Hellerstein MK. A dual sugar challenge test for lipogenic sensitivity to dietary fructose. J Clin Endocrinol Metab. 2011 Mar;96(3):861-8. doi: 10.1210/jc.2010-2007. Epub 2011 Jan 20. PMID 21252253
- [Background] Awai HI, Newton KP, Sirlin CB, Behling C, Schwimmer JB. Evidence and recommendations for imaging liver fat in children, based on systematic review. Clin Gastroenterol Hepatol. 2014 May;12(5):765-73. doi: 10.1016/j.cgh.2013.09.050. Epub 2013 Sep 30. PMID 24090729
- [Background] Shin HJ, Kim HG, Kim MJ, Koh H, Kim HY, Roh YH, Lee MJ. Normal range of hepatic fat fraction on dual- and triple-echo fat quantification MR in children. PLoS One. 2015 Feb 6;10(2):e0117480. doi: 10.1371/journal.pone.0117480. eCollection 2015. PMID 25659155
- [Background] Bonder A, Afdhal N. Utilization of FibroScan in clinical practice. Curr Gastroenterol Rep. 2014 Feb;16(2):372. doi: 10.1007/s11894-014-0372-6. PMID 24452634
- [Background] Lallukka S, Sadevirta S, Kallio MT, Luukkonen PK, Zhou Y, Hakkarainen A, Lundbom N, Orho-Melander M, Yki-Jarvinen H. Predictors of Liver Fat and Stiffness in Non-Alcoholic Fatty Liver Disease (NAFLD) - an 11-Year Prospective Study. Sci Rep. 2017 Nov 6;7(1):14561. doi: 10.1038/s41598-017-14706-0. PMID 29109528

RESULTS

PARTICIPANT FLOW:
Groups:
- High Genetic Risk Score (GRS) Group: This group consists of individuals who are in the highest quartile of the genetic risk score (GRS) and will ingest one sugar drink (equal to 2 soft drinks) per day for 3 weeks. The GRS is computed by adding the number of alleles that increase the risk for liver lipogenesis or fatty liver.
  Sugar drink: A sugar drink made with 1.2 g/kg body weight of added sugar( 0.75g/kg body weight of fructose + 0.45g/kg body weight of glucose) and 24oz water
- Low Genetic Risk Score (GRS) Group: This groups consists of individuals who are in the lowest quartile of the genetic risk score (GRS) and will ingest one sugar drink (equal to 2 soft drinks) per day for 3 weeks. The GRS is computed by adding the number of alleles that increase the risk for liver lipogenesis or fatty liver.
  Sugar drink: A sugar drink made with 1.2 g/kg body weight of added sugar( 0.75g/kg body weight of fructose + 0.45g/kg body weight of glucose) and 24oz water
Period: Overall Study
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Same as participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | High GRS Group | Low GRS Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.88 (9.6) | 24 (9.2) | 25.53 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Liver Fat Content Based on Elastography
Description: Elastography (Fibroscan) will be used to measure changes in liver fat.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | High GRS Group | Low GRS Group
Number analyzed (Participants) | 8 | 7
kilopascal (kPa) | -0.15 (0.85) | 1.10 (3.2)
Statistical Analysis 1: Comparison: High GRS Group vs Low GRS Group; The null hypothesis is that people with low GRS will have greater increase in liver fat as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.40, Paired t-test — All tests were individual tests; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.77 to 0.76], Standard Error of Mean 0.59

2. Primary Outcome: Mean Percent Change in Liver Fat Content Based on MRI
Description: Magnetic resonance imaging (MRI) will be used to measure changes in liver fat (% change in fat fraction).
Time Frame: between week 0 (Baseline) and week 3
Population: Due to COVID-19 limitations, only 4 participants had both the Week 0 (Baseline) and Week 3 MRIs.
Measure: Mean (Standard Deviation); unit: Percent fat fraction
Arm/Group | High GRS Group | Low GRS Group
Number analyzed (Participants) | 1 | 3
Percent fat fraction | -0.54 (0.00) | -0.33 (2.3)
Statistical Analysis 1: Comparison: High GRS Group vs Low GRS Group; The null hypothesis is that people with low GRS will have greater increase in liver fat as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.71, Paired t-test — All tests were individual tests; Mean Difference (Net) = -0.38, 95% CI 2-sided [-3.33 to 2.57], Standard Error of Mean 0.93

3. Primary Outcome: Mean Change in Serum Concentrations of Very Low Density Lipoprotein-triglycerides (VLDL-TG)
Description: VLDL-TG measurement in serum (mg/dl) at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg/dl | -0.021 (0.05) | -0.007 (0.03)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in VLDL-TG as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.0006, Paired t-test — All tests were individual tests; Mean Difference (Net) = -21.02, 95% CI 2-sided [-31.33 to -10.72], Standard Error of Mean 4.80

4. Primary Outcome: Mean Change in AUC of Serum Very Low Density Lipoprotein-triglycerides (VLDL-TG)
Description: Area under curve (AUC) (mg*hr/dl) of serum VLDL-TG for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg*hr/dl | 0.66 (0.35) | 0.75 (0.31)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; This analysis focuses on the changes in the area under the curve (AUC) for measurements at different time points between the two GRS groups; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.59, t-test, 2 sided; Median Difference (Net) = 0.094, 95% CI 2-sided [-0.27 to 0.46], Standard Error of Mean 0.17

5. Secondary Outcome: Mean Change in Serum Concentrations of Triglycerides
Description: Fasting concentrations of serum triglycerides (mg/dl) will be measured at week 0 and 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg/dl | 21.75 (60.6) | -2.14 (29.9)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in serum triglycerides as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.017, Paired t-test — All tests were individual tests; Mean Difference (Net) = -21.06, 95% CI 2-sided [-37.75 to -4.38], Standard Error of Mean 7.77

6. Secondary Outcome: Mean Change in AUC of Serum Triglycerides
Description: Area under curve (AUC) (mg*hr/dl) of serum VLDL-TG for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg*hr/dl | 0.59 (0.27) | 0.57 (0.35)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; This analysis focuses on the changes in the area under the curve (AUC) for measurements baseline and 3hr timepoints at week 0 and week 3 between the two GRS groups; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.89, t-test, 2 sided; Mean Difference (Net) = -0.022, 95% CI 2-sided [-0.37 to 0.33], Standard Error of Mean 0.16

7. Secondary Outcome: Mean Change in Serum Concentrations of HDL Cholesterol
Description: Fasting concentrations of serum HDL cholesterol (mg/dl) will be measured at week 0 and week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg/dl | -2.70 (15.9) | 0.39 (20.7)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have less increase in HDL cholesterol as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.36, Paired t-test — All tests were individual tests; Mean Difference (Net) = -4.36, 95% CI 2-sided [-14.28 to 5.55], Standard Error of Mean 4.62

8. Secondary Outcome: Mean Change in AUC of Serum HDL Cholesterol
Description: Area under curve (AUC) (mg*hr/dl) of serum HDL cholesterol for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg*hr/dl | 0.59 (0.30) | 0.66 (0.30)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.67, t-test, 2 sided; Mean Difference (Net) = 0.067, 95% CI 2-sided [-0.27 to 0.40], Standard Error of Mean 0.16

9. Secondary Outcome: Mean Change in Serum Concentrations of LDL Cholesterol
Description: Fasting concentrations of serum LDL cholesterol (mg/dl) will be measured.at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg/dl | -4.40 (36.2) | 0.96 (13.6)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in LDL cholesterol as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.09, Paired t-test — All tests were individual tests; Mean Difference (Net) = -21.03, 95% CI 2-sided [-45.76 to 3.69], Standard Error of Mean 11.53

10. Secondary Outcome: Mean Change in AUC of Serum LDL Cholesterol
Description: Area under curve (AUC) (mg*hr/dl) of serum LDL cholesterol for baseline and 3hr time points at week 0 and Week 3.
Time Frame: Week 0 (baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | High GRS Group | Low GRS Group
Number analyzed (Participants) | 8 | 7
mg*hr/dl | 0.63 (0.27) | 0.68 (0.25)
Statistical Analysis 1: Comparison: High GRS Group vs Low GRS Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.69, t-test, 2 sided; Mean Difference (Net) = 0.054, 95% CI 2-sided [-0.24 to 0.34], Standard Error of Mean 0.13

11. Secondary Outcome: Mean Change in Serum Concentrations of Total Cholesterol
Description: Fasting serum concentrations of total cholesterol (mg/dl) will be measured at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg/dl | -2.77 (53.2) | 0.92 (25.21)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in total cholesterol as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.07, Paired t-test — All tests were individual tests; Mean Difference (Net) = -29.61, 95% CI 2-sided [-62.39 to 3.17], Standard Error of Mean 15.28

12. Secondary Outcome: Mean Change in AUC of Serum Total Cholesterol
Description: Area under curve (AUC) (mg*hr/dl) of serum total cholesterol for baseline and 3hr time points at week 0 and Week 3.
Time Frame: week 0 and week 3
Population: Adolescent and young adults of Caucasian descent.
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
mg*hr/dl | 0.63 (0.27) | 0.66 (0.27)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.80, t-test, 2 sided; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.26 to 0.33], Standard Error of Mean 0.14

13. Secondary Outcome: Mean Changes in Serum Concentrations of Uric Acid
Description: Fasting concentrations of serum uric acid (ng/ml) will be measured at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
ng/ml | 0.21 (1.14) | -0.36 (0.89)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in serum uric acid as compared to high GRS group; Test type: Other; p = 0.17, Paired t-test — All tests were individual tests; Mean Difference (Net) = 0.36, 95% CI 2-sided [-0.18 to 0.91], Standard Error of Mean 0.25

14. Secondary Outcome: Mean Changes in AUC of Serum Uric Acid
Description: Area under curve (AUC) (ng*hr/ml) of serum uric acid for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
ng*hr/ml | 0.73 (0.27) | 0.52 (0.38)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.22, t-test, 2 sided; Mean Difference (Net) = -0.217, 95% CI 2-sided [-0.58 to 0.15], Standard Error of Mean 0.17

15. Secondary Outcome: Mean Change in Serum Concentrations of Liver Function Marker (Alanine Transaminase- ALT).
Description: Fasting concentrations of serum ALT (nmol) will be measured at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | High GRS Group | Low GRS Group
Number analyzed (Participants) | 8 | 7
nmol | -0.02 (0.05) | -0.007 (0.03)
Statistical Analysis 1: Comparison: High GRS Group vs Low GRS Group; The null hypothesis is that people with low GRS will have greater increase in serum ALT as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.04, Paired t-test — All tests were individual tests; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.03 to -0.0009], Standard Error of Mean 0.007

16. Secondary Outcome: Mean Change in AUC of Serum Alanine Transaminase (ALT)
Description: Area under curve (AUC) (nmol/hr) of serum ALT for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: nmol/hr
Arm/Group | High GRS Group | Low GRS Group
Number analyzed (Participants) | 8 | 7
nmol/hr | 0.66 (0.30) | 0.54 (0.42)
Statistical Analysis 1: Comparison: High GRS Group vs Low GRS Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.53, t-test, 2 sided; Mean Difference (Net) = -0.121, 95% CI 2-sided [-0.52 to 0.28], Standard Error of Mean 0.19

17. Secondary Outcome: Mean Change in Serum Concentrations of Liver Function Marker (Aspartate Transaminase-AST).
Description: Serum concentrations of serum AST will be measured at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
IU/L | -1.91 (14.9) | 1.28 (2.8)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in serum AST as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.25, Paired t-test — All tests were individual tests; Mean Difference (Net) = 20.57, 95% CI 2-sided [-16.9 to 58.08], Standard Error of Mean 17.5

18. Secondary Outcome: Mean Change in AUC of Serum Aspartate Transaminase (AST).
Description: Area under curve (AUC) (IU*hr/L) of serum AST for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: IU*hr/L
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
IU*hr/L | 0.61 (0.28) | 0.73 (0.17)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.20, t-test, 2 sided; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.59 to 0.13], Standard Error of Mean 0.17

19. Secondary Outcome: Mean Change in Serum Concentrations of Liver Function Marker (Alkaline Phosphatase-ALP)
Description: Fasting concentrations of serum ALP (nmol) will be measured at week 0 and week3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
nmol | 20.38 (71.14) | -5.24 (21.27)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in serum ALP as compared to high GRS group; Test type: Other; p = 0.21, Paired t-test — All tests were individual tests; Mean Difference (Net) = 28.95, 95% CI 2-sided [-17.76 to 75.67], Standard Error of Mean 21.78

20. Secondary Outcome: Mean Change in AUC of Serum Alkaline Phosphatase (ALP)
Description: Area under curve (AUC) (nmol/hr) of serum ALP for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: nmol/hr
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
nmol/hr | 0.63 (0.29) | 0.68 (0.16)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.67, t-test, 2 sided; Mean Difference (Net) = 0.054, 95% CI 2-sided [-0.214 to 0.321], Standard Error of Mean 0.12

21. Secondary Outcome: Mean Change in Serum Concentrations of Liver Function Marker (Gamma Glutamyl Transpeptidase-GGT)
Description: Serum concentrations of GGT will be measured at week 0 and week 3
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
IU/L | 0.26 (0.61) | 0.01 (0.04)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; The null hypothesis is that people with low GRS will have greater increase in serum GGT as compared to high GRS group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.41, Paired t-test — All tests were individual tests; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.12 to 0.28], Standard Error of Mean 0.09

22. Secondary Outcome: Mean Change in AUC of Serum Gamma Glutamyl Transpeptidase (GGT)
Description: Area under curve (AUC) (IU*hr/dl) of serum VLDL-TG for baseline and 3hr time points at week 0 and Week 3.
Time Frame: between week 0 (Baseline) and week 3
Population: Adolescents and young adults of Caucasian descent
Measure: Mean (Standard Deviation); unit: IU*hr/L
Arm/Group | High Genetic Risk Score (GRS) Group | Low Genetic Risk Score (GRS) Group
Number analyzed (Participants) | 8 | 7
IU*hr/L | 0.61 (0.31) | 0.50 (0.28)
Statistical Analysis 1: Comparison: High Genetic Risk Score (GRS) Group vs Low Genetic Risk Score (GRS) Group; Test type: Other — Both groups received the same intervention; however, their genetic make-up was different; p = 0.49, t-test, 2 sided; Mean Difference (Net) = -0.109, 95% CI 2-sided [-0.44 to 0.22], Standard Error of Mean 0.15

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through completion of study, a total of 3 weeks.
Arm/Group | High GRS Group | Low GRS Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03783195/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03783195/ICF_000.pdf